CLINICAL TRIAL: NCT00554632
Title: The Effects of Oral Contraceptive Pills vs Hormonal Patch on Coagulation Parameters
Brief Title: Birth Control Pill vs Birth Control Patch Study
Acronym: PvP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Vermont Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 03-168
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-10

CONDITIONS: Venous Thrombosis
Keywords: Contraceptive; Venous thrombosis; Coagulation parameter
MeSH Terms: conditions — Venous Thrombosis | interventions — norgestimate, ethinyl estradiol drug combination; Moxifloxacin; Ethinyl Estradiol; norelgestromin; Ortho Evra

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Use of transdermal hormonal contraceptive
  Interventions: Drug: Ethinyl estradiol and norelgestromin
- 2 (Active Comparator): Use of oral hormonal contraceptive
  Interventions: Drug: Ethinyl estradiol and norgestimate

INTERVENTIONS:
Drug: Ethinyl estradiol and norgestimate — Oral contraceptive
  Other Names: Ortho Cyclen
  Arms: 2
Drug: Ethinyl estradiol and norelgestromin — Transdermal hormonal contraceptive changed weekly
  Other Names: Ortho Evra
  Arms: 1

SUMMARY:
This study was a randomized, investigator-blinded, cross-over, clinic trial using twenty-four healthy women aged 18-35. All women received two months of the birth control patch or birth control pill, two months without any drug, then two months of the alternative drug. The birth control patch contained 0.75 milligrams ethinyl estradiol and 6 milligrams norelgestromin. The birth control pill contained 35 micrograms ethinyl estradiol and 250 micrograms norgestimate. Blood samples were taken before and after each treatment and were analyzed for the following lab values: D-dimer, von Willebrand factor, factor VIII, total and free protein S, antithrombin, fibrinogen, C-reactive protein and normalized activated protein C sensitivity ratio (nAPCsr). Two thrombin generation-based assays were used: the α2macroglobulin-thrombin endpoint method (α2M-IIa) and calibrated automated thrombinography (CAT).

DETAILED DESCRIPTION:
Twenty-four non-pregnant women 18-35 years of age, who had not been on hormonal contraception for at least 2 months prior to the study or who were least 3 months postpartum and non-lactating, were enrolled in this study between October 2003 and February 2005. The study protocol was approved by the University of Vermont Institutional Review Board, and all participants gave written informed consent. Exclusion criteria for participation were personal or family history of venous thromboembolism or coagulation disorders, pregnancy, uncontrolled hypertension, cardiovascular disease, complicated migraine headaches, breast cancer, diabetes, abnormal uterine bleeding, liver disease, or desire for pregnancy in less than 6 months.

This study was a randomized investigator-blind, cross-over clinical trial. The daily oral contraceptive contained 35 micrograms ethinyl estradiol and 250 micrograms norgestimate (Ortho Cylen®). The weekly transdermal hormonal contraceptive contained 0.75 milligrams ethinyl estradiol and 6.0 milligrams norelgestromin (Ortho Evra®). Norelgestromin is the active progestin metabolite of orally administered norgestimate. For the oral form the average steady state plasma concentration (Css) of ethinyl estradiol was 49.3 picograms/milliliter and of norelgestromin 0.73 nanograms/milliliter and for the transdermal form these concentrations were 80.0 picograms/milliliter and 0.888 nanograms/milliliter, respectively at the end of the second month of use.17 The average weekly exposure, calculated as area under the curve (AUC0-168pg.h/mL) for ethinyl estradiol was 55% higher with transdermal than with the oral contraceptive. The maximum ethinyl estradiol and norelgestromin levels (Cmax) were 133 pg/ml and 2.16 ng/ml for the oral form and 97.4 pg/ml and 1.12 ng/ml for the transdermal form.17 The application location of the patch does not alter the Css or Cmax.18 Medications were supplied to the patients by a research nurse and the completed packets were returned to document compliance. The contraceptives and the funding for the study were supplied by research grants from the University of Vermont Department of Obstetrics and Gynecology.

Prior to enrollment, participants underwent a physical examination including gynecologic examination. Women on hormonal contraceptives at recruitment were given barrier contraceptives for two months prior to starting the study. Participants were assigned a random identification number which indicated the sequence in which transdermal or oral contraceptives would be given. The daily oral contraceptive or weekly transdermal contraceptive was given with the typical dosing of three weeks active treatment followed by one week without hormone use. Following the first two months of hormonal contraceptive, each participated returned to barrier contraceptive for a two month washout period, then received two months of the alternative hormonal contraceptive. The investigators were blind to the order of contraceptive assigned for each participant.

There were four phlebotomies performed for each subject. Blood was drawn on menstrual cycle day 18 to 21 prior to the study, within 4 days of either the last pill or removal of the last patch, and on cycle day 18 to 21 in the second month of the washout period. Blood was collected using standardized methods with minimal stasis into vacutainer tubes, immediately placed on ice and centrifuged at 4oC. Plasma and serum was stored at -70oC until completion of the study.

Laboratory assays were performed in batch with each participant's serial samples analyzed in the same run. D-dimer, von Willebrand factor and antithrombin were measured using immuno-turbidometric assays on the STA-R analyzer (Liatest D-Di, Liatest vWF, Liatest ATIII, Diagnostica Stago, Parsippany, NJ) with coefficients of variation (CVs) of 3.0%, 3.85%, and 4.0-8.0% respectively. Factor VIII was determined by measuring the clotting time of the sample in factor VIII deficient plasma (STA-Deficient VIII; Diagnostica Stago, Parsippany, NJ) with a CV of 3.5%. Free and total protein S were measured by immunoassay (Asserachrom Free and Total Protein S, Diagnostica Stago, Parsippany, NJ) with CVs of 14.0% and 4.0% respectively. Fibrinogen and C-reactive protein were measured by immunonephelometry using the BNII instrument (N Antiserum to Human Fibrinogen, N High Sensitivity CRP, Dade-Behring, Deerfield, IL) with CVs of 2.3-4% and 2.6% respectively.

The normalized activated protein C sensitivity ratio (nAPCsr) was measured using two thrombin generation assays. In the first assay, coagulation was triggered in defibrinated plasma with tissue factor in the presence and absence of activated protein C and the amount of thrombin captured in complex with a2-macroglobulin over 30 minutes was taken as a measure for thrombin generation and used to calculate the nAPCsr (nAPCsr α2M-IIa).14 In the second assay, the nAPCsr (nAPCsr CAT) was determined by measuring thrombin generation in the presence and absence of activated protein C in full plasma in real-time with a fluorogenic thrombin substrate using calibrated automated thrombinography (CAT).19 The CV's of the nAPCsr α2M-IIa and nAPCsr CAT were 3.5% and 7%, respectively.

Repeated measures analyses of variance corresponding to a cross-over design incorporating both baseline and washout periods were used to determine the significance associated with differences between the hormonal contraceptive treatments for each of the biomarkers tested. Pre-planned contrasts were used to test for differences between the pre-treatment periods corresponding to oral and transdermal active treatments. Contrasts were also used to test for changes from pre-treatment to active treatment within each treatment and to determine whether these changes were parallel across the two active treatments. Biomarkers that had non-normal distributions based on residual plots were log transformed prior to analysis. Based on the analyses of variance results, there was no evidence of any significant order effects for any of the biomarkers. Analyses were performed using SAS Version 8.2 (SAS Institute, Cary, NC). Statistical significance was determined based on a=.05

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-35 years of age
* Not on hormones for at least 2 months prior to enrollment
* Must be more than 3 months post-partum, &
* Generally healthy.

Exclusion Criteria:

* Women with prior history of contraindications to taking birth control pills
* History of Deep Vein Thrombosis or Pulmonary Embolism
* Known history of coagulation disorders
* Liver disease
* Pregnant or actively attempting pregnancy
* Currently breastfeeding
* Uncontrolled hypertension
* Migraines with ischemic changes, &
* Weight more than 199 lbs.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-04; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change in coagulation parameters on transdermal versus oral contraceptive | 2003--2005

SECONDARY OUTCOMES:
Compare ethinyl estradiol levels for transdermal versus oral contraceptives | September 2007

CONTACTS AND LOCATIONS:
Overall Officials: Julia V Johnson, MD, Principal Investigator — Fletcher Allen Health Care & University of Vermont

REFERENCES:
- [Derived] Johnson JV, Lowell J, Badger GJ, Rosing J, Tchaikovski S, Cushman M. Effects of oral and transdermal hormonal contraception on vascular risk markers: a randomized controlled trial. Obstet Gynecol. 2008 Feb;111(2 Pt 1):278-84. doi: 10.1097/AOG.0b013e3181626d1b. PMID 18238963